CLINICAL TRIAL: NCT07236827
Title: A Comparison of Endoscopic Synchronous Injection and Submucosal Dissection(ESISD) and Conventional Endoscopic Submucosal Dissection(CESD) for Granular Mixed Nodular Laterally Spreading Tumor in the Rectum (LST-G-M)
Acronym: ESISD vs CESD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taihe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TaiheH
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Endoscopic Resection; Rectal Tumor
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Synchronous Injection and Submucosal Dissection (Experimental): Experimental group
  Interventions: Procedure: Endoscopic Synchronous Injection and Submucosal Dissection(ESISD)
- Conventional Endoscopic Submucosal Dissection (Active Comparator): compare group
  Interventions: Procedure: Conventional Endoscopic Submucosal Dissection(ESD)

INTERVENTIONS:
Procedure: Endoscopic Synchronous Injection and Submucosal Dissection(ESISD) — ESISD eliminates the need for injection needles or specialized submucosal agents by integrating injection and dissection into a single procedure. This approach reduces procedural costs, shortens the operation time, and enhances hemostasis during dissection. Additionally, it minimizes electrosurgical carbonization of the knife, preserving its cutting efficacy. The simplicity and broad applicability of ESISD can enhance traditional ESD workflows, warranting further validation across diverse patient populations.
  Other Names: Conventional Endoscopic Submucosal Dissection
  Arms: Endoscopic Synchronous Injection and Submucosal Dissection
Procedure: Conventional Endoscopic Submucosal Dissection(ESD) — ESD provides a minimally invasive approach for curative treatment of benign, precancerous, and early neoplastic lesions in the gastrointestinal tract
  Arms: Conventional Endoscopic Submucosal Dissection

SUMMARY:
What is the study about? This study introduces and evaluates a new endoscopic technique called Endoscopic Synchronized Injection and Submucosal Dissection (ESISD). It is designed to remove large, flat precancerous growths in the rectum, known as Granular Mixed Nodular Laterally Spreading Tumors (LST-G-M). We compared this new technique to the standard procedure, Conventional Endoscopic Submucosal Dissection (ESD), to see if it is safer, faster, and more efficient.

Who is this for? This research is intended for patients with large, flat rectal polyps, their families seeking the latest treatment options, and healthcare providers interested in advancements in minimally invasive gastroenterology procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Endoscopic diagnosis of a large (≥ 20 mm) granular mixed nodular laterally spreading tumor (LST-G-M) located in the rectum.
3. Lesion situated 0-15 cm from the anal verge.
4. Pre-procedure imaging (e.g., EUS) and endoscopic assessment suggest a very low to low risk of lymph node metastasis (i.e., lesions confined to the mucosa or with superficial submucosal invasion < 1000 μm).
5. Deemed suitable for Endoscopic Submucosal Dissection (ESD) based on a comprehensive clinical evaluation by the endoscopist.
6. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Coagulopathy that cannot be adequately corrected, including an international normalized ratio (INR) > 1.5 or a platelet count < 50,000/μL.
2. Evidence of deep submucosal invasion (≥ 1000 μm) or obvious non-lifting sign, suggesting a need for surgical intervention.
3. Pregnancy or lactation.
4. Inability to tolerate deep sedation or general anesthesia.
5. History of colorectal surgery (except for simple appendectomy or polypectomy).
6. Presence of a synchronous colorectal cancer that requires priority treatment.
7. Recurrent lesions at the same site.
8. Any condition that, in the investigator's opinion, could increase the patient's risk or interfere with the study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
procedure time | From enrollment to the end of treatment at 1 day
Hospitalization cost | From enrollment to the end of treatment at 10 days

SECONDARY OUTCOMES:
The rate of complete resection | From enrollment to the end of treatment at 1 day
The rate curative resection | From enrollment to the end of treatment at 10 days

IPD SHARING:
Plan to Share IPD: Undecided